CLINICAL TRIAL: NCT00872417
Title: Research on the Antiretroviral Therapy and Immune Reconstitution on Chinese HIV/AIDS Patients
Brief Title: Study on the Antiviral Therapy and Immune Reconstitution of Chinese HIV/AIDS Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Li Taisheng, MD, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CACT0810; PUMCH
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Acquired Immune Deficiency Syndrome; HIV Infections
Keywords: HIV/AIDS; antiretroviral therapy; immune reconstitution
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment-naive (Experimental): To explore the efficiency and safety of generic antiretroviral drugs for 520 treatment-naive HIV/AIDS patients
  Interventions: Drug: first line ARV (3TC+NVP+D4T or 3TC+NVP+AZT)
- TREATMENT-EXPERIENCED (No Intervention): To explore the long term ARV of treatment-experienced patients who have no sign of drug resistance; to explore the long term efficiency and safety and drug sife effects of ARV in HIV/AIDS patients. These patients have taken ARV for approximately 3 years already.
- drug resistance (Experimental): To explore the second line drugs for those drug resistance patients
  Interventions: Drug: second line ARV therapy (3TC+TDF+LPV/RTV)

INTERVENTIONS:
Drug: first line ARV (3TC+NVP+D4T or 3TC+NVP+AZT) — use the generic regimens: 3TC+NVP+D4T or 3TC+NVP+AZT to initiate the ARV therapy, after 6 months, half of the group 3TC+NVP+D4T patients switch to the the treatment of 3TC+NVP+AZT
  Arms: Treatment-naive
Drug: second line ARV therapy (3TC+TDF+LPV/RTV) — Use 3TC+TDF+LPV/RTV to treat those drug resistance patients, to explore the efficiency and safety of the second line ARV available in China
  Arms: drug resistance

SUMMARY:
This study will recruit 520 treatment-naive and 150 treatment-experienced patients to take the first line or second line of antiviral therapy. This study aims to set up a well-trained clinical and laboratory team in China, to explore the effects and side-effects of the first-line and the second line of ARV treatment in Chinese HIV/AIDS adult patients, to investigate the side-effects of ARV drugs, such as hepatotoxicity, lipoatrophy, cardiovascular influence, to explore the pharmacokinetics/pharmacodynamics (PK/PD) of Chinese generic ARV regiments and effective drug concentrations and to explore primary and secondary drug resistance in China and the immune reconstitution characters of long term ARV in Chinese adult AIDS patients. This study might provide more practical and optimizing prove for the treatment guideline for resource limited areas.

DETAILED DESCRIPTION:
Three arms will be studied in this research, 520 naive-treatment patients would be randomized to two groups, taking the generic drugs 3TC+D4T+NVP or AZT+3TC+NVP, 6 months later half of the 3TC+D4T+NVP group will switch to AZT+3TC+NVP, in order to observe the efficiency and safety of the first line drugs. Arm 2 will recruit 100 patients who are taking ARV for about three years already. Arm 3 will recruit 150 patients who have a Viral load of more than 1000 copies/ml, i.e., drug resistance. The second line drug 3TC+TDF+LPV/RTV will given to them and the safety and efficiency will be observed. All patients should be explored in terms of the clinical features, drugs side-effects, and immunological and viral response. The drug concentration and the metabolism changes would be explored also. Also the immune reconstitution will be studied for all patients. This study will be the first large-scale, multicentered, randomised, prospective ARV therapy study in China for HIV/AIDs patients. The result would provide proves for further practical antiviral therapy for China or other resource limited countries.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-65 years
* HIV seropositive and confirmed by western blot
* antiretroviral therapy naive for arm 1
* CD4 cell count < 350/mm3
* good adherence and follow up in the same place

Exclusion Criteria:

* pregnancy and breastfeeding
* AIDS defining illness or any infectious disease occured in one month but still unstable within 14 days
* with WBC < 2000/ul, neutrophil count < 1000/ul, hemoglobin < 9 g/dl, platelet count < 75000/ul, amylase > 2 ULN, transaminase or alkaline phosphatase or total bilirubin > 2 ULN, creatinine > 2 ULT.
* present acute or chronic pancreatitis
* intravenous drug user
* peripheral nephropathy
* severe nephropathy or mental disorder
* severe gastral ulcer
* heart or brain arthrosclerosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To set up a platform of antiviral therapy network all of CHINA, to obtain evidence to make first line or second line ARV treatment strategy for HIV/AIDS patients in resource limited areas. | two years

SECONDARY OUTCOMES:
Set up our own antiviral therapy guideline and drug side-effects, drug concentration and immune reconstitution result. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Tai sheng LI, M.D, Study Chair — PUMCH
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Fan H, Guo F, Hsieh E, Chen WT, Lv W, Han Y, Xie J, Li Y, Song X, Li T. Incidence of hypertension among persons living with HIV in China: a multicenter cohort study. BMC Public Health. 2020 Jun 1;20(1):834. doi: 10.1186/s12889-020-08586-9. PMID 32487185
- [Derived] Han Y, Li Y, Xie J, Qiu Z, Li Y, Song X, Zhu T, Li T. Week 120 efficacy of tenofovir, lamivudine and lopinavir/r-based second-line antiretroviral therapy in treatment-experienced HIV patients. PLoS One. 2015 Mar 30;10(3):e0120705. doi: 10.1371/journal.pone.0120705. eCollection 2015. PMID 25821963
- [Derived] Cao Y, Han Y, Xie J, Cui Q, Zhang L, Li Y, Li Y, Song X, Zhu T, Li T. Impact of a tenofovir disoproxil fumarate plus ritonavir-boosted protease inhibitor-based regimen on renal function in HIV-infected individuals: a prospective, multicenter study. BMC Infect Dis. 2013 Jul 1;13:301. doi: 10.1186/1471-2334-13-301. PMID 23815472
- [Derived] Kou H, Du X, Li Y, Xie J, Qiu Z, Ye M, Fu Q, Han Y, Zhu Z, Li T. Comparison of nevirapine plasma concentrations between lead-in and steady-state periods in Chinese HIV-infected patients. PLoS One. 2013;8(1):e52950. doi: 10.1371/journal.pone.0052950. Epub 2013 Jan 24. PMID 23359265
- [Derived] Wang H, Li Y, Zhang C, Han Y, Zhang X, Zhu T, Li T. Immunological and virological responses to cART in HIV/HBV co-infected patients from a multicenter cohort. AIDS. 2012 Sep 10;26(14):1755-63. doi: 10.1097/QAD.0b013e328355ced2. PMID 22614885